CLINICAL TRIAL: NCT06964789
Title: The Mechatronic Remote Physiotherapy System (MRPS) in Remote Stroke Rehabilitation: A Pilot Controlled Trial for 'Early Supported Discharge'
Brief Title: The Mechatronic Remote Physiotherapy System (MRPS) in Remote Stroke Rehabilitation
Acronym: MRPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Technology, Sligo (Other)
Collaborators: Sligo General Hospital (Other)
Responsible Party: Principal Investigator, Kenneth Monaghan, Director Kenneth Monaghan, Institute of Technology, Sligo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATU Sligo
Record Dates: First submitted 2024-10-23; First posted 2025-05-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Neurological Disorder
Keywords: Remote rehabilitation; Neurorehabilitation; Upper limb; Lower limb; Early Supported Discharge
MeSH Terms: conditions — Stroke; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Single blinded/masked design. As participants will be receiving either remote enhanced ESD or traditional therapist present ESD, blinding/masking of participants is not possible as they will be aware of the intervention they receive. Outcome measure assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants in the experimental group will receive enhanced ESD through the MRPS.
  The intervention will be given for approximately 6-8 weeks in total. Frequency will be determined by how often the participants' use the MRPS themselves. Frequency of use and level of completion of each session will be monitored. Enhanced ESD therapy sessions will be designed to reflect traditional ESD sessions.
  Interventions: Device: Mechatronic Remote Physiotherapy System (MRPS)
- Control (Active Comparator): Participants in the control group will receive traditional ESD. The intervention will be given for approximately 6-8 weeks in total with a frequency of 1-3 therapy visits per week (as per traditional ESD). Therapy sessions will be designed by therapists delivering the ESD service
  Interventions: Other: Early Supported Discharge

INTERVENTIONS:
Device: Mechatronic Remote Physiotherapy System (MRPS) — The MRPS is an Online Rehabilitation Platform for neurology patients. The platform has been designed to provide supervised and monitored remote rehabilitation therapy, initially focusing on patients who have suffered a stroke. The system comprises of a patent pending mirror therapy strengthening device, which is a neural therapy device using mirror therapy and exercise apparatus for upper limb rehabilitation. The platform also permits the addition of modules beneficial to the patients' recovery. A sensory substitution balance apparatus and motion detecting sensors are also being designed to connect to the system to allow for lower limb rehabilitation.
  Other Names: MRPS
  Arms: Experimental
Other: Early Supported Discharge — ESD is a multidisciplinary service providing medically stable patients continued therapy and healthcare in the community.
  Other Names: ESD
  Arms: Control

SUMMARY:
The aim of this pilot trial is to examine and compare the safety and feasibility of enhanced Early Supported Discharge (ESD) through the Mechatronic Remote Physiotherapy System (MRPS) and traditional ESD after stroke.

The main questions this trial aims to answer are:

* Is enhanced ESD via the MRPS safe, feasible and significantly different compared to traditional ESD when administered to patients after stroke?
* Do patients interact with and are they satisfied with the MRPS?
* Is enhanced ESD cost-effective compared to traditional ESD?
* Are there any adverse effects of the MRPS and what are the areas for further improvement?

Participants in the experimental group will receive enhanced ESD through the MRPS.

The intervention will be given for approximately 6-8 weeks in total. Frequency will be determined by how often the participants' use the MRPS themselves. Frequency of use and level of completion of each session will be monitored. Enhanced ESD therapy sessions will be designed to reflect traditional ESD sessions.

Participants in the control group will receive traditional ESD. The intervention will be given for approximately 6-8 weeks in total with a frequency of 1-3 therapy visits per week (as per traditional ESD). Therapy sessions will be designed by therapists delivering the ESD service.

DETAILED DESCRIPTION:
The Mechatronic Remote Physiotherapy System (MRPS) is an Online Rehabilitation Platform for neurology patients. The platform has been designed to provide supervised and monitored remote rehabilitation therapy, initially focusing on patients who have suffered a stroke. The system comprises of a patent pending mirror therapy strengthening device, which is a neural therapy device using mirror therapy and exercise apparatus for upper limb rehabilitation. The platform also permits the addition of modules beneficial to the patients' recovery. The use of a sensory substitution balance apparatus and motion capturing sensors are also being developed to allow for lower limb rehabilitation.

Participants will be randomly allocated to an experimental (n=7) or control group (n=7) using a block stratified randomization process. Block randomization will be stratified for age, gender and degree of disability (computer-generated random numbers) with allocation concealment.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of stroke;
* Completed inpatient rehabilitation;
* A level of ability that would allow them to participate safely (as determined by ESD team);
* Cognitive ability to consent and take part;
* Technological ability and resources to allow them to access MRPS platform;
* A proficiency in the English Language.

Exclusion Criteria:

* Involvement in other studies or rehabilitation programmes;
* A level of disability that would prevent them from participating safely (as determined by ESD team);
* Low level technological literacy or resources (e.g. Wi-Fi) which would prevent access to MRPS platform;
* Have uncontrolled medical condition or another serious medication condition in addition to stroke;
* Unable to understand or follow directions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Protocol Adherence/Compliance Rate. | through study completion, an average of 1 year
  Percentage of scheduled procedures, visits, or assessments completed as planned. 95% adherence/compliance rate suggest strong adherence/compliance rate.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS). | through study completion, an average of 1 year
  Outcome measure to assess static and dynamic balance with high validity and reliability within the stroke population. The Berg Balance Scale (BBS) is a clinical tool used to assess a person's balance through a series of 14 functional tasks, each scored on a scale from 0 to 4, with a maximum total score of 56. An increase in total BBS score from baseline indicates improved balance. A change of 6-7 points is often considered the minimal detectable change (MDC) in older adults or people with balance issues (i.e., change likely reflects a real improvement, not measurement error).
Fugl Meyer Assessment (FMA). | through study completion, an average of 1 year
  Stroke-specific, performance-based impairment index outcome measure. The Fugl-Meyer Assessment (FMA) is a widely used, validated tool to evaluate motor function, balance, sensation, and joint performance in individuals after a stroke. It is particularly focused on motor recovery and is considered one of the most comprehensive quantitative measures of physical impairment post-stroke. The full Fugl-Meyer Assessment includes 5 domains, with a total possible score of 226 points. Higher scores indicate better motor recovery/function. Change in score over time reflects improvement or decline.
  In stroke rehabilitation:10-point increase in motor score is typically considered clinically meaningful. Smaller changes (e.g., 5-7 points) may still be relevant depending on the baseline and context.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Monaghan, PhD, Study Director — ATU Sligo